CLINICAL TRIAL: NCT06106646
Title: Assessing the Effect of Vitamin C on Infant Lung Function When Given to Pregnant Women Who Smoke - (Long Term Follow-up of a Randomized Trial)
Brief Title: Vitamin C to Decrease Effects of Smoking in Pregnancy on Infant Lung Function (VCSIP) Longer Term Follow Up
Acronym: VCSIP
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Indiana University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Cynthia McEvoy, Principal Investigator, Oregon Health and Science University
Other Study IDs: VCSIP LTFU; R01HL162951 (NIH)
Record Dates: First submitted 2023-10-09; First posted 2023-10-30 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Asthma; Pulmonary Function; Wheezing; In Utero Nicotine
Keywords: Asthma; Pulmonary Function; Pulmonary Function Testing; Wheeze; Vitamin C; Antioxidants; Forced Expiratory Flows; Spirometry; Lung Function; Epigenetics; High resolution CT scans
MeSH Terms: conditions — Asthma; Respiratory Sounds

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — hair, buccal swabs, nasal swabs, blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Offspring of smokers who received Vitamin C: In the original VCSIP study, pregnant women were randomized to receive either extra Vitamin C every day (500mg/day) or placebo.
  Interventions: Dietary Supplement: No active intervention in this protocol (previously randomized to Vitamin C)
- Offspring of smokers who received Placebo: In the original VCSIP study, pregnant women were randomized to receive either extra Vitamin C every day (500mg/day) or placebo.
  Interventions: Other: No active intervention in this protocol (previously randomized to Placebo)
- Offspring of non-smokers

INTERVENTIONS:
Dietary Supplement: No active intervention in this protocol (previously randomized to Vitamin C) — In the original VCSIP study, pregnant women were randomized to receive either extra Vitamin C every day (500mg/day) or placebo. This trial is a follow-up trial with no active intervention.
  Groups: Offspring of smokers who received Vitamin C
Other: No active intervention in this protocol (previously randomized to Placebo) — In the original VCSIP study, pregnant women were randomized to receive either extra Vitamin C every day (500mg/day) or placebo. This trial is a follow-up trial with no active intervention.
  Groups: Offspring of smokers who received Placebo

SUMMARY:
The overall aims of this protocol are to determine whether prenatal supplementation with vitamin C to pregnant smokers can improve pulmonary function at 10 years of age in their offspring. This is an additional continuation of the Vitamin C to Decrease Effects of Smoking in Pregnancy on Infant Lung Function (VCSIP) trial, to follow the offspring through 10 years of age. The hypothesis for this protocol is an extension of the VCSIP trial that supplemental vitamin C in pregnant smokers can significantly improve their children's airway function tests. The investigators aim to demonstrate sustained improvement in airway/pulmonary function and trajectory through 10 years of age.

DETAILED DESCRIPTION:
The primary outcome of this longitudinal follow-up study is the comparison of airway function tests (specifically the forced expiratory flow between 25%and 75% of expired volume [FEF25-75]) measured yearly through 10 years of age by forced expiratory maneuvers with spirometry between the children of the pregnant smokers randomized to vitamin C (500 mg/day) versus placebo during pregnancy. The occurrence of wheeze obtained with quarterly standardized respiratory questionnaires will also be compared between the two groups of children. This is a follow-up of the original "Vitamin C to Decrease Effects of Smoking in Pregnancy on Infant Lung Function" (VCSIP) trial.

The secondary outcomes are:

1. A single low dose high-resolution computed tomography (HRCT) image of the lungs (acquired during inspiration) will be done at 10 years of age in offspring of pregnant smokers who were randomized to vitamin C (500 mg/day) versus placebo during pregnancy. Image analysis will be performed by Dr. Miranda Kirby's Quantitative Image Analysis in Medicine laboratory at Ryerson University in Toronto, ON using certified pulmonary image analysis software. The airway lumen cross sectional areas to at least the fifth generation of airways will be compared between the two groups of children. The number of airways and the lumen, wall, and total cross sectional areas and the segment lengths will also be quantified.
2. A secondary aim is to quantify the differences in DNA methylation between the two groups and measure the correlation between the differences in DNA methylation and respiratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women and their offspring randomized to vitamin C versus placebo during pregnancy as well as pregnant nonsmokers and their offspring enrolled as the reference group in the original VCSIP study

Exclusion Criteria:

* participants who specifically withdraw consent

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a follow up of NCT01723696. In that study, pregnant smokers were recruited at obstetric clinics delivering at OHSU in Portland OR, PeaceHealth Southwest Washington Medical Center in Vancouver, Washington or Indiana University in Indianapolis, Indiana. We are continuing to follow the offspring of those pregnant smokers (and control group non-smokers).
Sampling Method: Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Sustained improvement in pulmonary function and trajectory | 10 years of age
  The primary outcome of this longitudinal follow-up study is the comparison of airway function tests (specifically FEF25-75 in liters/sec) measured yearly through 10 years of age by forced expiratory maneuvers with spirometry between the children of the pregnant smokers randomized to vitamin C (500 mg/day) versus placebo during pregnancy. This is a follow-up of the original "Vitamin C to Decrease Effects of Smoking in Pregnancy on Infant Lung Function" (VCSIP) trial.

SECONDARY OUTCOMES:
Occurrence of wheeze | 10 years of age
  The occurrence of wheeze obtained with quarterly standardized respiratory questionnaires will also be compared between the children of the pregnant smokers randomized to vitamin C (500 mg/day) versus placebo during pregnancy. This is a follow-up of the original "Vitamin C to Decrease Effects of Smoking in Pregnancy on Infant Lung Function" (VCSIP) trial.
Airway lumen cross sectional areas | 10 years of age
  A single low dose high-resolution computed tomography (HRCT) image of the lungs (acquired during inspiration) will be done at 10 years of age in offspring of pregnant smokers who were randomized to vitamin C (500 mg/day) versus placebo during pregnancy. Image analysis will be performed by Dr. Miranda Kirby's Quantitative Image Analysis in Medicine laboratory at Ryerson University in Toronto, ON using certified pulmonary image analysis software. The airway lumen cross sectional areas (in mm squared) to at least the fifth generation of airways will be compared between the two groups of children.
Changes in DNA methylation | 10 years of age
  A secondary aim is to quantify the differences in DNA methylation between the two groups and measure the correlation between the differences in DNA methylation and respiratory outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy McEvoy, MD, MCR, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - Oregon Health and Science University (OHSU), Portland, Oregon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McEvoy CT, Schilling D, Clay N, Jackson K, Go MD, Spitale P, Bunten C, Leiva M, Gonzales D, Hollister-Smith J, Durand M, Frei B, Buist AS, Peters D, Morris CD, Spindel ER. Vitamin C supplementation for pregnant smoking women and pulmonary function in their newborn infants: a randomized clinical trial. JAMA. 2014 May;311(20):2074-82. doi: 10.1001/jama.2014.5217. PMID 24838476
- [Background] McEvoy CT, Shorey-Kendrick LE, Milner K, Harris J, Vuylsteke B, Cunningham M, Tiller C, Stewart J, Schilling D, Brownsberger J, Titus H, MacDonald KD, Gonzales D, Vu A, Park BS, Spindel ER, Morris CD, Tepper RS. Effect of Vitamin C Supplementation for Pregnant Smokers on Offspring Airway Function and Wheeze at Age 5 Years: Follow-up of a Randomized Clinical Trial. JAMA Pediatr. 2023 Jan 1;177(1):16-24. doi: 10.1001/jamapediatrics.2022.4401. PMID 36409489
- [Background] McEvoy CT, Shorey-Kendrick LE, Milner K, Schilling D, Tiller C, Vuylsteke B, Scherman A, Jackson K, Haas DM, Harris J, Park BS, Vu A, Kraemer DF, Gonzales D, Bunten C, Spindel ER, Morris CD, Tepper RS. Vitamin C to pregnant smokers persistently improves infant airway function to 12 months of age: a randomised trial. Eur Respir J. 2020 Dec 3;56(6):1902208. doi: 10.1183/13993003.02208-2019. Print 2020 Dec. PMID 32616589
- [Background] Blue SW, McEvoy CT, Spindel ER, Shorey-Kendrick LE, Davies MH, O'Sullivan SM, Erikson DW. Analysis of nicotine in plasma, brain, and hair samples with the same liquid chromatography-tandem mass spectrometry method. Rapid Commun Mass Spectrom. 2023 Sep 15;37(17):e9613. doi: 10.1002/rcm.9613. No abstract available. PMID 37580504
- [Background] McEvoy CT, Shorey-Kendrick LE, Milner K, Schilling D, Tiller C, Vuylsteke B, Scherman A, Jackson K, Haas DM, Harris J, Schuff R, Park BS, Vu A, Kraemer DF, Mitchell J, Metz J, Gonzales D, Bunten C, Spindel ER, Tepper RS, Morris CD. Oral Vitamin C (500 mg/d) to Pregnant Smokers Improves Infant Airway Function at 3 Months (VCSIP). A Randomized Trial. Am J Respir Crit Care Med. 2019 May 1;199(9):1139-1147. doi: 10.1164/rccm.201805-1011OC. PMID 30522343
- [Background] Shorey-Kendrick LE, McEvoy CT, O'Sullivan SM, Milner K, Vuylsteke B, Tepper RS, Haas DM, Park B, Gao L, Vu A, Morris CD, Spindel ER. Impact of vitamin C supplementation on placental DNA methylation changes related to maternal smoking: association with gene expression and respiratory outcomes. Clin Epigenetics. 2021 Sep 19;13(1):177. doi: 10.1186/s13148-021-01161-y. PMID 34538263